CLINICAL TRIAL: NCT06306768
Title: Remote Therapeutic Monitoring for Longitudinal Exercise and Self-Efficacy Tracking in Persons With Parkinson's Disease and Multiple Sclerosis.
Brief Title: Remote Therapeutic Monitoring Exercise Tracking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Miriam Rafferty, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00219979
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Multiple Sclerosis
Keywords: physical activity; exercise tracking; remote therapeutic monitoring; quality of life; self-efficacy
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote Therapeutic Monitoring (Other): Participants will receive 1 year of remote therapeutic monitoring via a connected health app and personal activity tracker to monitor their physical activity and exercise behaviors.
  Interventions: Device: Activity Monitoring

INTERVENTIONS:
Device: Activity Monitoring — Tracking participants step activity, workout frequency, minutes in target heart rate zone, and type of exercises completed over 1 year period. Goals will be set and customized by a research physical therapist to participants based on best practice recommendations.
  Other Names: Datos Health App

SUMMARY:
The purpose of this study is to examine physical activity and exercise behaviors in people with Parkinson's Disease and Multiple Sclerosis over the course of 1-year using a cloud-based remote monitoring platform.

DETAILED DESCRIPTION:
Remote therapeutic monitoring (RTM) is a reimbursable clinical service. Pilot investigation conducted by our lab demonstrated promise that this service is feasible to add to clinical care. It is unclear still if RTM is able to provide clinical benefit to patients including improving and sustaining physical activity (PA) and exercise behaviors over a longer period of time (>1 year). Our central hypothesis is that the addition of RTM to physical activity, both in a skilled rehabilitation program and within a home program, will improve long term outcomes related to physical activity including self-efficacy for exercise, consistent participation in home exercise recommendations, and quality of life in people living with PD and MS. Thus the specific aims of this study are as follows:

1. To assess PA and exercise behaviors over 1-year period using a remote therapeutic monitoring platform

   a. We will track steps per day, minutes of aerobic activity per week, and frequency of workouts including flexibility, balance, and resistance training.
2. To understand how engagement with RTM for PA tracking affects overall self-efficacy for exercise, readiness for exercise behavior change, and quality of life.

   1. Assessed through monthly self-report of usability survey for RTM and self-efficacy for exercise survey.

ELIGIBILITY:
Inclusion Criteria:

* Are ambulatory as their primary means of mobility without an assistive device except for single point cane or walking sticks in community
* Have a diagnosis of Parkinson's disease (Hoehn and Yahr 1-3), Parkinsonism, or Multiple Sclerosis
* Personal goal and willingness to address physical activity
* Have a smart phone (Datos Health app is compatible with any Smart phone device)
* Willing to accept Datos' Terms and Conditions

Exclusion Criteria:

* Individuals with cognitive or communication disorders (including dementia) which would limit their ability to interact with the RTM

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Metric 1 | Daily, through study completion, average 1 year
  steps per day
Physical Activity Metric 2 | Daily, through study completion, average 1 year
  Minutes of aerobic physical activity per day (moderate to vigorous physical activity)

SECONDARY OUTCOMES:
Exercise Self Efficacy | Completed every other month, through study completion, average of 1 year
  sums of 9 items with total scores ranging from 0-90; higher scores indicating higher self-efficacy.
Quality of Life from PROMIS 10-b | Completed every 3 months, through study completion, average of 1 year
  PROMIS 10-b short form which is 10 items measuring mobility difficulty, scores are summed and then translated to t-score.
Quality of Life from PROMIS-29 | Completed every 3 months, through study completion, average of 1 year
  PROMIS-29 measures seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and sleep disturbance).

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Rafferty, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Block VA, Pitsch E, Tahir P, Cree BA, Allen DD, Gelfand JM. Remote Physical Activity Monitoring in Neurological Disease: A Systematic Review. PLoS One. 2016 Apr 28;11(4):e0154335. doi: 10.1371/journal.pone.0154335. eCollection 2016. PMID 27124611
- [Background] Proschinger S, Kuhwand P, Rademacher A, Walzik D, Warnke C, Zimmer P, Joisten N. Fitness, physical activity, and exercise in multiple sclerosis: a systematic review on current evidence for interactions with disease activity and progression. J Neurol. 2022 Jun;269(6):2922-2940. doi: 10.1007/s00415-021-10935-6. Epub 2022 Jan 27. PMID 35084560
- [Background] Speelman AD, van de Warrenburg BP, van Nimwegen M, Petzinger GM, Munneke M, Bloem BR. How might physical activity benefit patients with Parkinson disease? Nat Rev Neurol. 2011 Jul 12;7(9):528-34. doi: 10.1038/nrneurol.2011.107. PMID 21750523